CLINICAL TRIAL: NCT01315535
Title: Evaluation of the Efficacy and Side Effects of Fast Mandibular Advancement With Oral Appliance in the Treatment of Obstructive Sleep Apnea Syndrome
Brief Title: Fast Titration of Oral Appliance at Obstructive Sleep Apnea Syndrome (OSAS) Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Associacao Fundo de Incentivo a Psicofarmcologia (Other)
Responsible Party: BITTENCOURT, LIA R. A. / PhD, UNIFESP
Other Study IDs: CEP0301/10
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-03

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Mandibular Advancement; Oral Appliance; TMD
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Fast Titration
- Regular Titration
- Fast Tritation Including Mandibular Exercises
- Regular Tritation Including Mandibular Exercises

SUMMARY:
The literature does not discuss if the fast oral appliance titration (30 days period) in Obstructive Sleep Apnea Syndrome (OSAS) treatment, may improve subjects quality of life in such brief period. Temporomandibular dysfunction-related (TMD) is one of the most important side effects observed in OSAS treatment with oral appliance. Since the effectiveness of mandibular exercises in the control of TMD pain has already been verified, it may play a fundamental role in the support of the fast oral appliance titration.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 35kg/m2
* MILD TO MODERATE OSAS DIAGNOSIS ACCORDING TO THE AASM CRITERIA (2005)
* Negative TMD diagnosis (according to RDC/TMD)

Exclusion Criteria:

* DENTAL CONDITIONS THAT CONTRAINDICATED THE ORAL APLLIANCE USAGE
* SLEEP DISORDERS OTHER THAN OSAS

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with mild to moderate osas, according to the aasm criteria (2005) from the respiratory disorders clinic (UNIFESP) referred to oral appliance treatment.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Do Sono / Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil